CLINICAL TRIAL: NCT06667999
Title: The Intensive Care Platform Trial (INCEPT)
Brief Title: The Intensive Care Platform Trial
Acronym: INCEPT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Anders Perner (Other)
Collaborators: Rigshospitalet, Denmark (Other); Bispebjerg Hospital (Other); Herlev Hospital (Other); Hillerod Hospital, Denmark (Other); Kolding Sygehus (Other); Zealand University Hospital (Other); Slagelse Hospital (Other); Viborg Regional Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other); Gødstrup Hospital (Other); Copenhagen University Hospital, Hvidovre (Other); Odense University Hospital (Other); Randers Regional Hospital (Other); University of Copenhagen (Other); North Denmark Region (Other Government); Region Capital Denmark (Other); Region Zealand (Other); University Medical Center Groningen (Other); Steno Diabetes Center Copenhagen (Other); Karolinska Institutet (Other); Oslo University Hospital (Other); University Hospital, Basel, Switzerland (Other); Tampere University (Other); Collaboration of Research in Intensive Care (Unknown); Danish Intensive Care Database (Unknown); The National University Hospital of Iceland (Unknown)
Responsible Party: Sponsor-Investigator, Anders Perner, Professor, senior staff specialist, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RH-ITA-2024-516208-41-00; 2024-516208-41-00 (EU CTIS Number); U1111-1313-8171 (Other: World Health Organization - Universal Trial Number)
Record Dates: First submitted 2024-10-25; First posted 2024-10-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Intensive Care Patients; Intensive Care Unit Patients; Critical Illness
Keywords: Platform trial; Intensive care; Intensive care unit; Critical illness; Clinical platform trial
MeSH Terms: conditions — Critical Illness | interventions — Albumins; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: Randomised, embedded, multifactorial, adaptive, primarily Bayesian, domain-based platform trial.
Masking Description: Domains may be open-label or blinded (masked). Outcome assessment of health-related quality of life and cognitive function will always be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Albumin (Experimental): Use of albumin in ICU during circulatory failure in addition to crystalloids (resuscitation) and for substitution in case of suspected or overt albumin loss or plasma albumin levels ≤25 g/L
  Interventions: Drug: Albumin
- No albumin use (Other): No albumin is to be used in ICU unless specific events occur
  Interventions: Other: No albumin use
- Low-molecular-weight heparin for thromboprophylaxis in weight-adjusted dose (Experimental): Use of low-molecular-weight heparin for thromboprophylaxis in weight-adjusted dose during ICU stay
  Interventions: Drug: LMWH in weight-adjusted dose
- Low-molecular-weight heparin for thromboprophylaxis in fixed low dose (Active Comparator): Use of low-molecular-weight heparin for thromboprophylaxis in fixed low dose during ICU stay
  Interventions: Drug: LMWH in fixed low dose
- Low-molecular-weight heparin for thromboprophylaxis in fixed intermediate dose (Active Comparator): Use of low-molecular-weight heparin for thromboprophylaxis in fixed intermediate dose during ICU stay
  Interventions: Drug: LMWH in fixed intermediate dose

INTERVENTIONS:
Drug: Albumin — Albumin should be used for the following indications: 1. During circulatory failure in addition to crystalloids (resuscitation). 2. For substitution in case of: suspected or overt albumin loss OR P-albumin levels below or equal to 25 g/L. Decisions around timing, volume, and concentration of albumin, and its use for other indications, are at the clinician's discretion. P-albumin should be measured according to local practice.
  Arms: Albumin
Other: No albumin use — Albumin should not be used. In case of the following special circumstances, albumin may be considered: 1. Large ascites drainage (i.e., equal to or more than 1 L tapped) 2. Spontaneous bacterial peritonitis 3. Hepatorenal syndrome.
  Arms: No albumin use
Drug: LMWH in weight-adjusted dose — Patients with indication for thromboprophylaxis receive low-molecular-weight heparin (LMWH) in a weight-adjusted dose during their ICU stay. The treating clinician may decide to adjust or withhold one or more doses in case of acute and/or chronic kidney injury, renal replacement therapy, thrombocytopenia, invasive procedures, use of thrombolysis, and active (major) bleeding.
  Arms: Low-molecular-weight heparin for thromboprophylaxis in weight-adjusted dose
Drug: LMWH in fixed low dose — Patients with indication for thromboprophylaxis receive low-molecular-weight heparin (LMWH) in a fixed low dose during their ICU stay. The treating clinician may decide to adjust or withhold one or more doses in case of acute and/or chronic kidney injury, renal replacement therapy, thrombocytopenia, invasive procedures, use of thrombolysis, and active (major) bleeding.
  Arms: Low-molecular-weight heparin for thromboprophylaxis in fixed low dose
Drug: LMWH in fixed intermediate dose — Patients with indication for thromboprophylaxis receive low-molecular-weight heparin (LMWH) in a fixed intermediate dose during their ICU stay. The treating clinician may decide to adjust or withhold one or more doses in case of acute and/or chronic kidney injury, renal replacement therapy, thrombocytopenia, invasive procedures, use of thrombolysis, and active (major) bleeding.
  Arms: Low-molecular-weight heparin for thromboprophylaxis in fixed intermediate dose

SUMMARY:
Among critically ill patients, many die, and many of the survivors and their family members struggle for years with reduced quality of life. Critically ill patients are treated in intensive care units (ICUs). Here, they receive life support, e.g., mechanical ventilation and advanced support of the circulation (heart and blood vessels) and kidneys. In addition, ICU patients receive many other treatments. It is, however, uncertain if all the treatments provide value for the patients. The desirable effects of many treatments are uncertain, and some may be wasteful or even harmful.

Clinical trials are necessary to validly assess the desirable and undesirable effects of different treatments. However, conventional clinical trials have limitations:

* They typically only assess a single question related to a single comparison of treatments at a time.
* They are often not very flexible, including with regards to the number of participants needed, and this increases the risk that a trial will end up as inconclusive.
* There is no or limited re-use or sharing of infrastructure across trials, leading to duplicate work and resource use.
* Trial participants do usually not benefit from the obtained knowledge before the trial concludes.
* Involvement of patients, family members, and other stakeholders is typically limited, which may decrease the relevance of the questions addressed.

With the Intensive Care Platform Trial (INCEPT), we aim to tackle these challenges by establishing a flexible platform trial that continuously learns from the obtained results. The platform trial may run forever with simultaneous and continuous assessment of many treatments. INCEPT will continuously learn from the accrued data and use these to improve the treatment of both participating and future patients. With INCEPT, we are also building a framework for thorough and extensive involvement of key stakeholders, including patients and family members. INCEPT will improve the way clinical trials are done and increase the probabilities that treatments are improved. This will:

* Directly improve outcomes for ICU patients.
* Relieve a strained healthcare system by discarding inefficient or harmful treatments.
* Ensure that new treatments are beneficial or cost-effective before implementation.
* Lower the costs and burdens of assessing more treatments in the critically ill.

DETAILED DESCRIPTION:
Background:

Randomised clinical trials (RCTs) are the gold standard for evaluating intervention effects, however, conventional RCTs are bureaucratic, costly, inflexible, and often inconclusive. Adaptive platform trials are increasingly used as they can reduce barriers and are more flexible, and thus come with a higher probability of obtaining conclusive results faster at lower costs.

Objectives:

The Intensive Care Platform Trial (INCEPT) will be used to assess the effects of interventions used in adults acutely admitted to the intensive care unit (ICU).

Design:

INCEPT is an investigator-initiated, pragmatic, randomised, embedded, multifactorial, international, adaptive platform trial. INCEPT uses adaptive stopping and arm-dropping rules, as well as fixed and response-adaptive randomisation. Specific domains may be either open label or blinded.

Domains and interventions:

Comparable groups of interventions will be nested in domains, which have conceptual similarities with stand-alone randomised trials. Domains will continuously be added to INCEPT and conducted following domain-specific appendices to the core protocol.

Inclusion and exclusion criteria:

Adults acutely admitted to the ICU will be screened if they are eligible for at least one active domain. The only platform-level exclusion criteria are 1) informed consent after inclusion expected to be unobtainable and 2) patients admitted under coercive measures. Additional inclusion and exclusion criteria will be domain-specific.

Stakeholder involvement:

Stakeholder involvement is central in INCEPT and ensured through a central advisory board comprising various key stakeholders, and consultations with national and international research panels consisting of ICU survivors, family members, clinicians, and researchers. Stakeholders will be involved in the development of the overall platform trial and specific domains with pre-specified minimum requirements for involvement.

Outcomes:

Each domain will use one of the core outcomes (defined elsewhere in the registration) as the primary outcome and the guiding outcome driving all adaptations.

Statistical methods Primary analyses will generally be conducted in the intention-to-treat population of each domain. INCEPT primarily uses Bayesian statistical methods with neutral priors conveying either minimal information or some scepticism, although specific domains may use conventional, frequentist statistical methods. Outcomes will generally be analysed using logistic and linear regression models adjusted for pre-specified anticipated prognostic baseline characteristics, followed by calculation of sample-average estimates and intervention effects using G-computation. Results will be presented for each intervention and comparisons presented on both the absolute (risk differences and mean differences) and relative (risk ratios and ratios of means) scales with 95% credible intervals and probabilities of superiority. INCEPT will generally use constant, symmetric stopping rules for superiority/inferiority based on the guiding outcome; domains may use stopping rules for practical equivalence or futility based on the posterior distribution of the guiding outcome on the absolute scale. All stopping rules will be binding. Response-adaptive randomisation, either with or without restrictions, may be used based on the posterior distribution for the guiding outcome. Missing data will be multiply imputed. Additional secondary analyses (e.g., per-protocol analyses), sensitivity analyses, and analyses of heterogeneity in intervention effects according to pre-defined baseline characteristics may be specified for each domain and undertaken once a domain has stopped. Domains will be designed and evaluated using statistical simulation.

ELIGIBILITY:
The general eligibility criteria below apply to INCEPT as a whole and thus to all domains. Domains may impose domain-specific eligibility criteria that restrict the population eligible for that domain further, but domains are not allowed to broaden the general eligibility criteria. Domain-specific eligibility criteria always apply to all arms in a domain.

PLATFORM INCLUSION CRITERIA:

* Adult patient (≥18 years old) acutely admitted to the ICU. This includes ICU admissions after emergency surgery, unplanned ICU admissions after elective surgery, and prolonged ICU admissions due to complications after elective surgery (i.e., admissions occurring or being prolonged due to an unexpected, worsened condition, but excluding planned ICU admissions after elective surgery without clinical deterioration).
* Eligible for at least one active domain.

PLATFORM EXCLUSION CRITERIA:

* Informed consent following inclusion expected to be unobtainable (e.g., known previous objections to participation).
* Patient is under coercive measures (e.g., ongoing involuntary hospital stay or under the jurisdiction of correctional authorities).

Patients who have previously been included in INCEPT may only be included again during new ICU admissions but may only be randomised to domains in which they have not previously been randomised.

DOMAIN-SPECIFIC ELIGIBLE CRITERIA:

Each domain may have additional eligibility criteria. Refer to the study website for more information (www.incept.dk).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
One of the INCEPT core outcomes (varying between domains) | From randomisation to 30-180 days after randomisation.
  Each domain in INCEPT will use one of the core outcomes; 1. All-cause 30-day mortality. 2. All-cause 90-day mortality. 3. All-cause 180-day mortality. 4. Days alive without life support at day 30. 5. Days alive without life support at day 90. 6. Days alive out of hospital at day 30. 7. Days alive out of hospital at day 90. 8. Days free of delirium at day 30. 9. EQ VAS (Health-Related Quality of Life) at day 180. 10. EQ-5D-5L index values (Health-related quality of life) at day 180. 11. Cognitive function at day 180 (all described under "secondary outcomes").
Days alive without life support at day 30 (Albumin domain) | From randomisation to 30 days after randomisation.
  Days alive without the use of life support, with life support defined as invasive mechanical ventilation (≥1 hour of ventilation through a cuffed tube), continuous (i.e., ≥1 hour) use of vasopressors/inotropes, use of renal replacement therapy (including any form of in-hospital renal replacement therapy [e.g., haemodialysis, haemofiltration, or haemodiafiltration], continuously or intermittently, and including days in between intermittent renal replacement therapy; pauses between renal replacement therapy of up to three days will be considered as days receiving intermittent renal replacement therapy) at hospitals. Integer (0-30 overall; 0-29 in domains with life support at baseline as an eligibility criterion).
Days alive and out of hospital at day 30 (Thromboprophylaxis domain) | From randomisation to 30 days after randomisation.
  Days alive and out of hospital. Rehabilitation facilities and nursing homes do not count as hospitals. Integer 0-29.

SECONDARY OUTCOMES:
All-cause 30-day mortality | 30 days after randomisation.
  All-cause, fixed-time mortality. Binary.
All-cause 90-day mortality | 90 days after randomisation.
  All-cause, fixed-time mortality. Binary.
All-cause 180-day mortality | 180 days after randomisation.
  All-cause, fixed-time mortality. Binary.
Days alive without life support at day 30 | From randomisation to 30 days after randomisation.
  Days alive without the use of life support, with life support defined as invasive mechanical ventilation (≥1 hour of ventilation through a cuffed tube), continuous (i.e., ≥1 hour) use of vasopressors/inotropes, use of renal replacement therapy (including any form of in-hospital renal replacement therapy [e.g., haemodialysis, haemofiltration, or haemodiafiltration], continuously or intermittently, and including days in between intermittent renal replacement therapy; pauses between renal replacement therapy of up to three days will be considered as days receiving intermittent renal replacement therapy) at hospitals. Integer (0-30 overall; 0-29 in domains with life support at baseline as an eligibility criterion).
Days alive without life support at day 90 | From randomisation to 90 days after randomisation.
  Days alive without the use of life support, with life support defined as invasive mechanical ventilation (≥1 hour of ventilation through a cuffed tube), continuous (i.e., ≥1 hour) use of vasopressors/inotropes, use of renal replacement therapy (including any form of in-hospital renal replacement therapy [e.g., haemodialysis, haemofiltration, or haemodiafiltration], continuously or intermittently, and including days in between intermittent renal replacement therapy; pauses between renal replacement therapy of up to three days will be considered as days receiving intermittent renal replacement therapy) at hospitals. Integer (0-90 overall; 0-89 in domains with life support at baseline as an eligibility criterion).
Days alive out of hospital at day 30 | From randomisation to 30 days after randomisation.
  Days alive and out of hospital. Rehabilitation facilities and nursing homes do not count as hospitals. Integer 0-29.
Days alive out of hospital at day 90 | From randomisation to 90 days after randomisation.
  Days alive and out of hospital. Rehabilitation facilities and nursing homes do not count as hospitals. Integer 0-89.
Days free of delirium at day 30 | From randomisation to 30 days after randomisation.
  Days free of delirium. Days are not considered free of delirium in case of any of the following: a) any registered positive delirium score with a validated screening tool (Confusion Assessment Method for the Intensive Care Unit [CAM-ICU], CAM-ICU-7 or Intensive Care Delirium Screening Checklist [ICDSC]) b) new treatment with antipsychotics (any administration of haloperidol, olanzapine, or quetiapine in participants not receiving either of these at the time of index hospital admission) c) delirium status not evaluable due to mortality or registered coma. Integer (0-30 overall; 0-29 in domains with delirium at baseline as an eligibility criterion).
EQ-5D-5L index values (Health-Related Quality of Life) at day 180 | 180 days after randomisation (+/- 14 days).
  EQ-5D-5L instrument with responses across five domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with five response levels each. Used with a value set to calculate index values anchored at 1 (perfect health) and 0 (a health state considered as bad as being dead) with index values below 0 representing health states worse than death. Preferably completed by participants, but completed by proxies if participants are unable to answer (using the proxy-participant perspective, i.e., the proxy will answer from the participant's perspective as the limited, indirect data available indicates that this perspective may better correspond to the participant's own response, if available). Decimal number (minimum values depend on value sets used, e.g., -0.758 with the Danish value set; maximum value: 1.000).
EQ VAS (Health-Related Quality of Life) at day 180 | 180 days after randomisation (+/- 14 days).
  A visual analogue scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state), part of the EQ-5D-5L instrument
Cognitive function at day 180 | 180 days after randomisation (+/- 14 days).
  Montreal Cognitive Assessment test 5-minute version, v2.1 ("Mini MoCA"), ranging from 0 points (worst) to 15 points (best).
Thromboprophylaxis domain specific secondary outcomes | 30 days (matching the primary and guiding outcome) and 90 days (matching the maximum intervention period).
  The number of participants with one or more domain-specific secondary outcomes, i.e., venous thromboembolism or major bleeding as specified in the domain-specific appendix.

OTHER OUTCOMES:
Albumin domain-specific safety outcomes | 30 days (matching the primary and guiding outcome) and 90 days (matching the maximum intervention period.
  Albumin domain: The number of participants with one or more safety outcomes, i.e. severe anaphylatic reaction or major bleedings as specified in the domain specific appendix.
Thromboprophylaxis domain-specific safety outcomes | 30 days (matching the primary and guiding outcome) and 90 days (matching the maximum intervention period).
  The number of participants with one or more safety outcomes, i.e. severe anaphylactic reaction to LMWH or heparin-induced thrombocytopenia as specified in the domain specific appendix.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, Professor, Study Chair — Copenhagen University Hospital - Rigshospitalet, Department of Intensive Care; Anders Granholm, MD, Principal Investigator — Copenhagen University Hospital - Rigshospitalet, Department of Intensive Care; Morten H Moeller, Professor, Principal Investigator — Copenhagen University Hospital - Rigshospitalet, Department of Intensive Care
Locations (21):
- Denmark (21):
  - Anaesthesia, Hospital Sønderjylland, Aabenraa
  - Department of Anaesthesia and Intensive Care, Aalborg University Hospital, Aalborg
  - Department of Intensive Care Nord , Aarhus University Hospital, Aarhus
  - Department of Intensive Care Øst, Aarhus University Hospital, Aarhus
  - Department of Cardiothoracic Anaesthesia and Intensive care, Copenhagen Universisty Hospital - Rigshospitalet, Copenhagen
  - Department of Intensive Care, Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Neuroanaesthesiology, Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Department of anesthesiology and intensive care, Bispebjerg-Frederiksberg Hospital, Copenhagen
  - Esbjerg Hospital, Esbjerg
  - Department of Anesthesiology and Intensive Care, Copenhagen University Hospital Herlev, Herlev
  - Department of Anaesthesiology and Intensive Care, Gødstrup Hospital, Herning
  - Department of Anaesthesia and Intensive Care Medicine, Copenhagen University Hospital - North Zealand, Hillerød
  - Anaesthesiology and Intensive Care, Amager and Hvidovre Hospital, Hvidovre
  - Department of Anesthesia and intensive care medicine, Kolding Hospital, Kolding
  - Department of Anesthesia, Zealand University Hospital, Køge
  - Anesthesiology (ICU), Zealand University Hospital, Nykøbing Falster, Nykøbing Falster
  - Department of Anesthesiology and Intensive Care, Odense University Hospital, Odense
  - Operation og Intensiv, Regional Hospital Randers, Randers
  - Intensive care, Slagelse Hospital, Slagelse
  - Department. of Anesthesiology and Intensive Care Medicine, Svendborg
  - Department of Anaesthesiology and Intensive Care, Regional Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: Yes
An anonymised version of the final dataset (without personal, identifiable information, with timestamps replaced by relative time differences with respect to the time of randomisation, and other measures as deemed relevant) in each domain may be shared with other researchers following a reasonable request (i.e., a research proposal outlining the objectives, methodologies, and plans for data usage) and subsequent approval by the platform and domain management committees. Any sharing of data that is not considered anonymised will be after the necessary approvals; alternatively, aggregation, scrambling, or synthetic datasets (i.e., datasets with similar structure and attempts to preserve the overall relationships between variables as the original dataset) may be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For each domain, data will generally only be shared after a grace period of at least 9 months following initial publication of results based on the data. Approved researchers will sign appropriate agreements to ensure compliance with the approved purpose and ethical and eventual legal requirements.
Access Criteria: Described in the core protocol which will be available at www.incept.dk once the trial has been approved.
URL: https://incept.dk

REFERENCES:
- See also: Trial website - core protocol and domain-specific appendices will be made available here once approved. — https://www.incept.dk